CLINICAL TRIAL: NCT03165708
Title: Identification of the Epidural Space: a Double Blind Comparison Between th CompuFlo® Epidural Computer Controlled System and the Standard LOR to Saline Technique in Obstetrics
Brief Title: Epidural Computer Controlled System for the Epidural Space Verification
Status: Completed | Type: Observational
Sponsor: Città di Roma Hospital (Other)
Responsible Party: Principal Investigator, Giorgio Capogna, Head Department Anesthesia, Città di Roma Hospital
Other Study IDs: 001
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Epidural
Keywords: Epidural technique

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anesthesiologist: The active comparators for this study will be expert anaesthesiologists (operator). The operators will be blinded to all visual and audible CompuFlo® real-time pressure feedbacks.Inter-rater agreement, or concordance, between an expert anaesthesiologist and the CompuFlo® Epidural Computer Controlled System for the epidural space verification will be assessed by blinded tagging of the operator's feeling of the ligamenta and epidural space on the screen of the Compuflo to be eventually compared with the pressure's variations

SUMMARY:
The purpose of this study will be to evaluate the inter-rater agreement, or concordance, between an expert anaesthesiologist and the CompuFlo® Epidural Computer Controlled System for the epidural space verification.

Primary study endpoint will be successful concordance of identification of ligamentum flavum and epidural space during a standard epidural procedure in pregnant patient. Secondary outcome will be successful concordance of identification of bony contact during a standard epidural procedure in pregnant patient.

DETAILED DESCRIPTION:
After skin local anesthesia and after the subcutaneous insertion of the epidural Tuohy needle, an independent investigator will make the O point of the CompuFlo® device that will be connected, via a three way stopcock, to the Tuohy needle in order to register, in a double blind way, the delta of pressures encountered by the needle during its advancement.

When the operator will reach the supraspinous ligament, a slight resistance will be encountered due to the nature of the bevel, and the density of the ligament. As soon as this resistance will be felt, the operator immediately will tell the investigator who will flag the CompuFlo® device. If no sensation will be felt the operator will tell "none" to the investigator.

The needle will be then advanced through the loose interspinous ligament which typically offers much less resistance than the sopraspinous ligament (often felt as a "no resistance feeling" in the obstetric patient). Once again, as soon as this loss or reduced or no resistance sensation is felt, the operator immediately will tell the investigator who will flag the CompuFlo® device. If no sensation will be felt the operator will tell "none" to the investigator.

According to the standard epidural technique, the point of the needle will be further advanced. The feeling of a greater increase of resistance, often associated with a "crunch", usually indicates the initial penetration of the needle in the rear wall of the ligamentum flavum. As soon as this resistance or "crunch" is felt, the operator immediately will tell the investigator who will flag the CompuFlo® device.

Then, the operator will remove the stylet and gently will attach to the needle a disposable 10 mL loss of resistance syringe containing a few millimeters (5-7 mL) of sterile saline solution and will open the three way stopcock in order to record both the pressures given-and-received by the CompuFlo® and the pressure produced by the operator's hand.

Constant, unremitting pressure will be now exerted on the plunger of the syringe by the thumb of the dominant hand of the operator in order to obtain the needle advancement solely by means of the pressure exerted by the operator on the plunger of the syringe.

As the point of the needle will emerge from the ligamentum flavum into the epidural space, the resistance suddenly will disappear and the advancement of the needle immediately will stop, (since the driving force exerted on the piston is discharged by the sudden entering of the liquid in the epidural space). As soon as this loss of resistance is felt, the operator immediately will tell the investigator who will who will flag the CompuFlo® device. The operator will stop the procedure for at least 10 seconds to allow the investigator to record the static epidural pressures.

ELIGIBILITY:
Inclusion Criteria:

* Parturients undergoing epidural block for cesarean section or labor analgesia

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy parturients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
concordance between anesthesiologist and Compuflo | during epidural technique performance
  Primary study endpoint will be successful concordance of identification of ligamentum flavum and epidural space during a standard epidural procedure in pregnant patient.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, Principal Investigator — Citta di Roma Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghelber O, Gebhard RE, Vora S, Hagberg CA, Szmuk P. Identification of the epidural space using pressure measurement with the compuflo injection pump--a pilot study. Reg Anesth Pain Med. 2008 Jul-Aug;33(4):346-52. doi: 10.1016/j.rapm.2008.01.012. PMID 18675746